CLINICAL TRIAL: NCT06637228
Title: Effects of Integrated Exercise on Sarcopenia, Depression Symptoms, and Quality of Life of Community-Dwelling Older Adults With Dementia
Brief Title: Effects of Integrated Exercise on Sarcopenia, Depression Symptoms, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: Tungs' Taichung Metroharbor Hospital (Unknown)
Responsible Party: Principal Investigator, Yu-Nu Wang, Associate Professor, Chang Gung University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZRRPF3N0031; TTMHH-R1130034 (Other Grant/Funding Number: Tungs' Taichung Metroharbor Hospital)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dementia; Depressive Symptoms; Quality of Life (QOL); Sarcopenia in Elderly
Keywords: dementia; older adults; sarcopenia; depression symptoms; quality of life; integrated exercise; cognitive function; geriatric care; health outcomes
MeSH Terms: conditions — Dementia; Depression; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment model, consisting of two groups: an integrated exercise intervention group and a control group. Participants aged 65 years and older with a diagnosis of dementia were recruited from outpatient neurological/dementia clinics and community centers in Taiwan. The intervention group engaged in a 12-week structured exercise program that included strength training, aerobic exercise, stretching, and balance activities, meeting at least three times per week. In contrast, the control group continued their usual daily activities without any structured exercise regimen. Both groups were assessed at baseline and post-intervention to evaluate the effects of the integrated exercise on sarcopenia, depression symptoms, and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group engaged in a structured integrated exercise program designed to improve physical function and emotional well-being. The program lasted for 12 weeks, with sessions held three times a week. Each session lasted for 50 minutes and included a combination of strength training, aerobic exercises, stretching, and balance activities. The exercise regimen aimed to enhance muscle strength, endurance, flexibility, and overall quality of life, specifically targeting the symptoms of sarcopenia and depression.
  Interventions: Behavioral: Move Your Hands, Feet, and Brain: Integrated Exercise Intervention Based on Taipei City Elderly Physical Activity Guidelines
- Control Group (No Intervention): The control group continued with their usual treatment and daily activities.

INTERVENTIONS:
Behavioral: Move Your Hands, Feet, and Brain: Integrated Exercise Intervention Based on Taipei City Elderly Physical Activity Guidelines — This video is tailored for fitness exercises for both healthy and sub-healthy elderly individuals and features various physical activity themes, including warm-up routines, balance and coordination drills, aerobic coordination exercises, strength training using chairs and water bottles, and cool-down routines. We selected a 3-month duration with sessions held three times a week to align with established effective intervention periods and to ensure participant adherence.
  Integrated exercise sessions were conducted by the staff at the dementia care centers/service bases and lasted 50 minutes. Considering the impact of dementia and aging on the ability of older adults to engage in physical activities, the staff provided simple instructions, and participants performed the exercises while seated to prevent falls. Meanwhile, the control group continued with their usual treatment and daily activities.
  Arms: Intervention Group

SUMMARY:
The goal of this quasi-experimental (nonrandomized intervention) study is to investigate the effects of an integrated exercise intervention on sarcopenia, depression symptoms, and quality of life in community-dwelling older adults with dementia. The main questions it aims to answer are:

1. Does the integrated exercise intervention improve muscle mass and strength in older adults with dementia?
2. How does the intervention affect the participants' depression symptoms?
3. What changes occur in the quality of life of participants following the exercise program?

In this study, participants will:

1. Be divided into two groups: an integrated exercise group and a control group.
2. The intervention group will participate in a 12-week integrated exercise program consisting of strength training, aerobic exercise, stretching, and balance training, performed for 50 minutes at least three times a week.
3. Assessments will be conducted before the intervention and after 12 weeks, including body composition analysis, grip strength measurement, physical function tests, and structured questionnaires evaluating demographics, depression symptoms, and quality of life.

This study aims to determine the effectiveness of integrated exercise in addressing sarcopenia, alleviating depression symptoms, and enhancing the quality of life among older adults with dementia. The findings may provide valuable insights for developing community-based exercise interventions for this population.

DETAILED DESCRIPTION:
This study explored the effects of an integrated exercise intervention on sarcopenia, depressive symptoms, and quality of life in community-dwelling older adults diagnosed with dementia. Sarcopenia, characterized by the loss of muscle mass and strength associated with aging, poses significant risks, including frailty, disability, and reduced quality of life, particularly among older adults.

Given the rising prevalence of dementia globally, addressing the effects of sarcopenia in this population was crucial. The proposed intervention involved a carefully structured exercise program tailored to enhance physical function and emotional health, incorporating elements of strength training, aerobic exercise, stretching, and balance activities.

Participants were recruited from outpatient neurological/dementia clinics and community centers in Taiwan, targeting individuals aged 65 and above. Selection was based on established eligibility criteria. Those assigned to the integrated exercise group engaged in a 12-week program, attending exercise sessions lasting 50 minutes at least three times per week. Meanwhile, the control group continued with their regular daily activities without any structured exercise regimen.

To assess the intervention's effectiveness, various outcome measures were utilized. These included evaluations of body composition, grip strength, and physical function, along with structured questionnaires to assess depressive symptoms and overall quality of life. Assessments took place at baseline and at the conclusion of the 12-week program, allowing for a comparison of pre- and post-intervention outcomes.

The findings from this study provided valuable insights into the role of structured physical activity in mitigating the effects of sarcopenia and enhancing mental health among older adults living with dementia. Ultimately, the results will inform the development of effective, community-based strategies aimed at improving the overall well-being of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Older adults with dementia were eligible to enroll in the study if they met the following inclusion criteria: 1) age of 65 years or older, 2) diagnosed with dementia by a neurologist, 3) able to walk independently (with or without a cane), 4) having measurable grip strength on at least one hand, 5) and having a score on the Clinical Dementia Rating (CDR) scale ≤ 2.

Exclusion Criteria:

* Individuals at risk of falling, unable to communicate or complete the sarcopenia test, under guardianship, any major psychiatric disorder, or any cognitive disability or impairment that prevented meaningful communication were excluded.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Sarcopenia Improvement | Baseline Assessment: 0 weeks (Pre-intervention); Post-Intervention Assessment: 12 weeks (Post-intervention)
  Participants were assessed for skeletal muscle mass, based on the skeletal muscle index (SMI), muscle strength, and physical performance using thresholds established by the AWGS to identify those with sarcopenia and group them as follows: possible sarcopenia (low muscle strength or low physical performance, only); sarcopenia (low SMI, and low muscle strength or low physical performance); and severe sarcopenia (low SMI, and low muscle strength, and low physical performance).

SECONDARY OUTCOMES:
Depression Symptoms | Baseline Assessment: 0 weeks (Pre-intervention); Post-Intervention Assessment: 12 weeks (Post-intervention)
  We used the Chinese version of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D), validated by Cheng & Chan (2005). This scale measures the frequency of depressive symptoms over the past week, with responses ranging from 0 (less than 1 day) to 3 (5-7 days). Total scores range from 0 to 60, with higher scores indicating more severe depressive symptoms.
Quality of Life | Baseline Assessment: 0 weeks (Pre-intervention); Post-Intervention Assessment: 12 weeks (Post-intervention)
  We used the Taiwan version of the Medical Outcomes Study Short Form-36 (SF-36) scale (Tseng, et al., 2003) to assess quality of life, which follows a norm-based scoring method (Ware et al., 1994) and Taiwan-specific algorithms. Scores range from 0 to 100, with higher scores indicating better QoL.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Dementia Care Center, Tungs' Taichung Metroharbor Hospital, Taichung
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Escriche-Escuder A, Fuentes-Abolafio IJ, Roldan-Jimenez C, Cuesta-Vargas AI. Effects of exercise on muscle mass, strength, and physical performance in older adults with sarcopenia: A systematic review and meta-analysis according to the EWGSOP criteria. Exp Gerontol. 2021 Aug;151:111420. doi: 10.1016/j.exger.2021.111420. Epub 2021 May 23. PMID 34029642
- [Result] Silva AC, Pereira MA, Peixoto LM, Rosse IC, Junior JBF, de Oliveira EC, Becker LK, Coelho DB. 12 weeks of resistance training with progressive intensity improves the diagnostic parameters of sarcopenia in individuals of advanced age. Geriatr Nurs. 2023 Nov-Dec;54:60-65. doi: 10.1016/j.gerinurse.2023.08.015. Epub 2023 Sep 11. PMID 37703691
- [Result] Gonzalez-Rocha A, Mendez-Sanchez L, Ortiz-Rodriguez MA, Denova-Gutierrez E. Effect Of Exercise on Muscle Mass, Fat Mass, Bone Mass, Muscular Strength and Physical Performance in Community Dwelling Older Adults: Systematic Review and Meta-Analysis. Aging Dis. 2022 Oct 1;13(5):1421-1435. doi: 10.14336/AD.2022.0215. eCollection 2022 Oct 1. PMID 36186132
- [Result] Lin A, Wang T, Li C, Pu F, Abdelrahman Z, Jin M, Yang Z, Zhang L, Cao X, Sun K, Hou T, Liu Z, Chen L, Chen Z. Association of Sarcopenia with Cognitive Function and Dementia Risk Score: A National Prospective Cohort Study. Metabolites. 2023 Feb 8;13(2):245. doi: 10.3390/metabo13020245. PMID 36837864
- [Result] Wang LT, Huang WC, Hung YC, Park JH. Association between Depressive Symptoms and Risk of Sarcopenia in Taiwanese Older Adults. J Nutr Health Aging. 2021;25(6):790-794. doi: 10.1007/s12603-021-1631-5. PMID 34179935
- [Result] Barros D, Borges-Machado F, Silva-Fernandes A, Ribeiro O, Carvalho J. Do physical fitness and cognitive function mediate the relationship between basic activities of daily living and quality of life in older adults with dementia? Qual Life Res. 2024 Apr;33(4):917-926. doi: 10.1007/s11136-023-03570-3. Epub 2023 Dec 19. PMID 38112863
- [Result] Beaudart C, Demonceau C, Reginster JY, Locquet M, Cesari M, Cruz Jentoft AJ, Bruyere O. Sarcopenia and health-related quality of life: A systematic review and meta-analysis. J Cachexia Sarcopenia Muscle. 2023 Jun;14(3):1228-1243. doi: 10.1002/jcsm.13243. Epub 2023 May 4. PMID 37139947
- [Result] Faieta JM, Devos H, Vaduvathiriyan P, York MK, Erickson KI, Hirsch MA, Downer BG, van Wegen EEH, Wong DC, Philippou E, Negm A, Ahmadnezhad P, Krishnan S, Kahya M, Sood P, Heyn PC. Exercise interventions for older adults with Alzheimer's disease: a systematic review and meta-analysis protocol. Syst Rev. 2021 Jan 4;10(1):6. doi: 10.1186/s13643-020-01555-8. PMID 33397453
- [Result] Liu W, Zhang J, Wang Y, Li J, Chang J, Jia Q. Effect of Physical Exercise on Cognitive Function of Alzheimer's Disease Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trial. Front Psychiatry. 2022 Jun 16;13:927128. doi: 10.3389/fpsyt.2022.927128. eCollection 2022. PMID 35782450
- [Result] Yoo SZ, No MH, Heo JW, Park DH, Kang JH, Kim SH, Kwak HB. Role of exercise in age-related sarcopenia. J Exerc Rehabil. 2018 Aug 24;14(4):551-558. doi: 10.12965/jer.1836268.134. eCollection 2018 Aug. PMID 30276173
- [Result] Shen Y, Shi Q, Nong K, Li S, Yue J, Huang J, Dong B, Beauchamp M, Hao Q. Exercise for sarcopenia in older people: A systematic review and network meta-analysis. J Cachexia Sarcopenia Muscle. 2023 Jun;14(3):1199-1211. doi: 10.1002/jcsm.13225. Epub 2023 Apr 14. PMID 37057640